CLINICAL TRIAL: NCT00352989
Title: Efficacy of Diosmectite (SMECTA®) in Combination With Oral Rehydration in the Treatment of Acute Watery Diarrhoea in Infants and Children. A Phase IIIB, Placebo Controlled, Randomized, Double Blind, Parallel Groups, Multicenter Study.
Brief Title: Effectiveness of Smecta in Combination With Oral Rehydration in the Treatment of Acute Watery Diarrhoea in Infants and Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-31-00250-101
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Diarrhoea
MeSH Terms: conditions — Diarrhea | interventions — smecta; Smectite; Duration of Therapy

INTERVENTIONS:
Drug: Smecta (Diosmectite), duration of treatment - 7 days

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Smecta at decreasing stool weight, when compared to placebo, in the treatment of acute diarrhoea in children.

ELIGIBILITY:
Inclusion Criteria:

* male
* acute watery diarrhoea defined as at least 3 watery stools per 24 hours
* duration of watery diarrhoea of less than 72 hours and with at least 1 watery stool for the last 12 hours
* dehydration signs requiring oral rehydration according to current WHO guidelines

Exclusion Criteria:

* severe dehydration that needs IV therapy
* presence of gross blood in stools
* fever >39 degrees Celsius

Ages: 1 Month to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2006-07; Primary Completion 2007-03-24 (Actual); Study Completion 2007-03-24 (Actual)

PRIMARY OUTCOMES:
Cumulative faecal output (g/kg of body weight) | 72 hours after first study drug intake

SECONDARY OUTCOMES:
Cumulative faecal output (g) | 72 hours after the first study drug intake
Faecal output (g/kg of body weight) per day | 72 hours after the first study drug intake
Duration of watery diarrhoea (time of first study drug intake to watery diarrhoea disappearance) | 7 days after the first study drug intake
Percentage of children withdrawn from the study due to IV rehydration (according to WHO guideline) | 7 days after the first study drug intake
Percentage of body weight gain in comparison with body weight at inclusion | Till 7 days after the first study drug intake
Percentage of children with at least one formed stool (H12, H24, H36, H48, H60, H72, then daily until Day 7) | Till 7 days after first study drug intake
Daily until Day 7: stool frequency, watery stool number, formed stool number, soft stool number, percentage of patients with bottom skin irritation, percentage of patients with anal irritation, appetite on a 100mm visual analogue scale | Till 7 days after first study drug intake
Tolerance of Smecta (assessed via adverse event reporting) | Till 7 days after the last study drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (19):
- Malaysia (19):
  - Kluang Hospital, Kluang, Johor
  - Kajang Hospital, Jalan Semenyih, Kajang
  - Kulim Hospital, Jalan Mahang, Kedah
  - Temerloh Hospital, Hospital Sultan Haji Ahmad Shah, Pahang
  - Seri Manjung Hospital, Seri Manjung, Perak
  - Teluk Intan Hospital, Teluk Intan, Perak
  - Alor Setar Hospital, Alor Setar Kedah
  - Ipoh Hospital, Ipoh - Perak
  - Raja Perempuan Zainab II Hospital, Kelantan
  - Tengku Ampuan Rahimah Hospital, Kuala Selangor
  - Serdang Hospital, Kuala Selangor
  - Kuala Terengganu Hospital, Kuala Terengganu
  - Tengku Ampuan Afzan Hospital, Kuantan Pahang
  - Sarawak General Hospital, Kuching
  - Malacca Hospital, Malacca
  - Tuanku Jaafar Hospital, Negeri Sembilan
  - Pulau Pinang Hospital, Pulau Pinang
  - Sungai Petani Hospital, Sungai Petani
  - Taiping Hospital, Taiping Perak